CLINICAL TRIAL: NCT05645874
Title: Reference Values of Intraepidermal Nerve Fiber Density in Children and Small Fiber Neuropathy in Children With Acquired and Genetic Neurodevelopmental Disorders - An Unrecognized Cause of Pain and Window Into Brain Pathology ? -
Brief Title: Reference Values of Intraepidermal Nerve Fiber Density in Children and Small Fiber Neuropathy in Neurodevelopmental Disorders
Acronym: SFN_children
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: SFN children; 2021-1556 (Other: Ethical review board - Medical faculty, Heinrich-Heine University, University Hospital Düsseldorf)
Record Dates: First submitted 2022-11-30; First posted 2022-12-12 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-03

CONDITIONS: Mitochondrial Diseases; Developmental Delay Disorder; Small Fiber Neuropathy; Cerebral Palsy
MeSH Terms: conditions — Mitochondrial Diseases; Developmental Disabilities; Small Fiber Neuropathy; Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Skin biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control (no underlying neurological disorder): Neurologically healthy individuals undergoing elective surgical intervention on the leg
  Interventions: Diagnostic Test: Skin biopsy
- Neurodevelopmental disorder_Genetic cause known: Individuals with neurodevelopmental symptoms (developmental delay, muscular hypotonia, seizures, ataxia, etc) with age of onset before the age of 18 years. Genetic etiology, if a genetic diagnosis had been established before inclusion to the study
  Interventions: Diagnostic Test: Skin biopsy
- Neurodevelopmental disorder_Acquird (cause known): Individuals with neurodevelopmental symptoms (developmental delay, muscular hypotonia, seizures, ataxia, etc) with age of onset before the age of 18 years.
  Acquired etiology, if a plausible cause of NDD was known (including but not limited to perinatal asphyxia, postnatal asphyxia or cardiopulmonary resuscitation, premature birth with periventricular leukomalacia, premature birth with severe intracranial bleeding, brain damage due to encephalitis, stroke, cerebral tumor; no red flags of genetic disease, such as syndromic features),
  Interventions: Diagnostic Test: Skin biopsy
- Neurodevelopmental disorder_Unexplained etiology: Individuals with neurodevelopmental symptoms (developmental delay, muscular hypotonia, seizures, ataxia, etc) with age of onset before the age of 18 years.
  Unexplained etiology, if there is no genetic diagnosis established so far and if there is no history of perinatal risk factors for brain injury or if there are other red flags for genetic cause (e.g., normal magnetic resonance findings or delayed myelination; findings suggestive of syndromic disease).
  Interventions: Diagnostic Test: Skin biopsy

INTERVENTIONS:
Diagnostic Test: Skin biopsy — Control skin biopsies from children without a chronic underlying disease are drawn from surgical crop margins during elective orthopedic surgery of the lower leg (n<80). Skin punch biopsies from children with acquired (n<80) or genetic NDD (n<80) or unknown etiology (N<80) are drawn in the setting of elective interventions during sedation or after local anesthesia. IENFD is quantified by immunohistochemistry and compared between the control and NDD group.

SUMMARY:
Background: Small-Fiber-Neuropathy describes the degeneration of mildly or unmyelinated nerve fibers and causes neuropathic pain and autonomic dysfunction. Gold standard for the diagnosis is a small skin punch biopsy from the lower leg and the histological quantification of the intraepidermal nerve fiber density (IENFD). In children, the normal IENFD has not been systematically assessed and normal reference values are needed. In Parkinson´s disease, the neurodegeneration also affects the peripheral nerves and SFN is present already in the early stages. Whether neurodevelopmental disorders (NDDs) in childhood are likewise associated with SFN is largely unknown. The IENFD is age-dependent and declines with age.

Aims: In this study, we are establishing the reference values for the physiological IENFD in children from 0-18 years. Moreover, we are investigating if children with NDDs have a reduced IENFD and if SFN is a clinically relevant cause of pain and autonomic dysfunction.

DETAILED DESCRIPTION:
In the first part of the study, skin biopsies will be collected from the leg from children with a normal neurological development (healthy children) in the setting of elective orthopedic surgery (during general anesthesia; from surgical crop margins).

The IENFD is determined by staining and quantification of PGP9.5-positive intraepidermal nerve fibers on 40 µm thick skin sections.

The skin biopsies will be collected from the site of orthopedic surgical procedure. For example, if the child is undergoing corrective osteotomy of genu valgum, the skin biopsy is drawn from the most distal part of surgical incision sides (distal leg); if the child is undergoing orthopedic surgery in the context of epiphyseolysis capitis femoris, the skin biopsy is drawn from the thigh (proximal leg):

In adults, the IENFD is higher in specimens derived from the proximal leg than in skin from the distal leg. Because in small fiber neuropathy the small nerve fiber degeneration often starts distally, the recommended sampling site for the quantification of IENFD in adults is the distal leg. That is why the calculation of the 5th percentile as the cutoff for reduced IENFD in children will be based on skin biopsies collected from the distal leg.

Due to the limited number of surgeries on the distal leg and distal biopsies in certain age groups of healthy participants (e.g. 4-8), cases with skin biopsies taken from the proximal leg will also be included. The IENFD from cases drawn from the proximal leg and cases from the distal leg will be compared. The samples drawn from the distal or proximal leg will be labelled accordingly. If the IENFD is comparable between the distal and proximal cases, a pooled analysis including proximal and distal cases will be performed.

In the second part of the study, skin biopsies from the distal leg will be collected from children with neurodevelopmental disorders of acquired, genetic and initially unexplained etiology in the setting of local anesthesia, whenever possible during an elective intervention with sedation/general anesthesia. IENFD below the predicted age- and sex-specific 5th percentile will be classified "reduced", otherwise as "normal".

A literature review will be performed to identify those neurodevelopmental disorders that have been associated with peripheral neuropathy in the past.

In cases with a yet unexplained etiology of neurodevelopmental disorder (no perinatal asphyxia, postnatal asphyxia, no cardiopulmonary resuscitation, no extreme prematurity, no encephalitis others, no stroke, or cerebral tumor), genetic testing (exome or genome sequencing and microarray analysis) will be performed.

Clinical symptoms of SFN (distal sensory signs and autonomic dysfunction) In adults the diagnosis of SNF is also based on the presence of distal sensory signs. Therefore, all participants or their legal guardians will be requested to answer questionnaires [(SFN-symptom inventory questionnaire (SFN-SIQ) and the SFN-Screening list (SFNSL)] that specifically assess distal sensory and autonomic symptoms related to SFN.

Additional exploratory subgroup analysis 1): In adults the diagnosis of SNF is also based on abnormal thermal perception assessed by quantitative sensory testing (QST). In collaboration with the University Children´s Hospital of the Ruhr University Bochum, QST will be performed in those children that are old enough and who have the cognitive ability to undergo QST. Small nerve fiber function including thermal perception will be assessed.

Additional exploratory subgroup analysis 2): Small fiber neuropathy can be associated with large fiber neuropathy. Therefore, the proportion of abnormal findings of electrophysiological studies in medical record of children with a reduced versus normal IENFD will be assessed.

ELIGIBILITY:
control patients

Inclusion Criteria:

* Elective surgical intervention from lower leg
* Interest to participate in the study, informed consent
* Unremarkable neurological development

Exclusion Criteria:

* Clinical signs of polyneuropathy, autonomic dysfunction
* Skin inflammation, scar, skin disease, other known chronic diseases that can cause small fiber pathology

Neurodevelopmental patients

Inclusion Criteria:

* Neurodevelopmental problems (developmental delay, muscular hypotonia, seizures, ataxia,...) with age of onset before the age of 18 years
* Interest to participate in the study, informed consent

Exclusion Criteria:

* Known polyneuropathy
* Skin inflammation, scar, skin disease, other known chronic diseases that can cause small fiber pathology

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. Control (no underlying neurological disorder) individuals
  2. Neurodevelopmental disorder_Genetic cause known
  3. Neurodevelopmental disorder_Acquired (cause known, for example perinatal asphyxia or intracranial bleeding)
  4. Neurodevelopmental disorder_Cause unknown
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Part 1 - Cutoff for reduced intraepidermal nerve fiber density (IENFD) in children | 2 years
  Age- and sex-specific 5th percentile of IENFD in the distal leg of neurologically healthy children aged 0-18 years (controls) as the cutoff for reduced IENFD.
Part 2 - Proportion of children with reduced IENFD among children with neurodevelopmental disorders (NDDs). | 2 years
  Proportion of children with genetic, acquired NDDs or NDDs of initially unexplained etiology whose IENFD falls below the predicted, age- and sex-specific 5th percentile (cutoff) that was calculated in part 1.

CONTACTS AND LOCATIONS:
Overall Officials: Felix Distelmaier, Principal Investigator — Department of General Pediatrics, Heinrich-Heine-University, Düsseldorf, Germany.
Locations (1):
- University Hospital Düsseldord, Department of General Pediatrics, Neonatology and Pediatric Cardiology, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After publication
Access Criteria: Email to principal investigators explaining why it might be helpful to share the data.

REFERENCES:
- [Background] Lauria G, Bakkers M, Schmitz C, Lombardi R, Penza P, Devigili G, Smith AG, Hsieh ST, Mellgren SI, Umapathi T, Ziegler D, Faber CG, Merkies IS. Intraepidermal nerve fiber density at the distal leg: a worldwide normative reference study. J Peripher Nerv Syst. 2010 Sep;15(3):202-7. doi: 10.1111/j.1529-8027.2010.00271.x. PMID 21040142